CLINICAL TRIAL: NCT03538977
Title: Effects of Hydrotherapy in Premature Infants With Bronchopulmonary Dysplasia During Hospitalization: a Randomized Clinical Trial
Brief Title: Hydrotherapy in Premature Infants With Bronchopulmonary Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Vanessa Suziane Probst, Principal investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEL-PPG Reabilitação
Record Dates: First submitted 2018-04-10; First posted 2018-05-29 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Hydrotherapy; Electromyography; Pain; Prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Pain; Premature Birth | interventions — Hydrotherapy; Baths

STUDY DESIGN:
Intervention Model Description: PTNB with a diagnosis of BPD will be randomized into two groups: conventional physiotherapy (GP) and conventional physiotherapy plus hydrotherapy (GH). The PTNB randomized to GH will be submitted to 11 hydrotherapy sessions. The PTNB from both groups will be submitted to evaluation of heart rate (HR), peripheral oxygen saturation (SpO2), respiratory rate (RR), pain, respiratory distress, sleep state, and wakefulness. The level of salivary cortisol and muscular activity (EMG) will also be evaluated.
Who Masked: Outcomes Assessor
Masking Description: For the evaluation of pain, respiratory effort and state of sleep and wakefulness, specific scales previously validated for this population will be used: NIPS (Neonatal Infant Pain Scale) scale, Silverman Andersen respiratory severity score, and the Brazelton Neonatal Behavioral Assessment Scale, respectively. Patients will be filmed during the five moments of assessment, and two physiotherapists blinded to the groups will watch the filming and perform the evaluation using the scales previously mentioned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy (GP) (Active Comparator): The sample will be evaluated once a day in the morning until they complete at least 11 intervention sessions of conventional physiotherapy in five moments: immediately before therapy, immediately after, 15, 30 and 60 minutes after the intervention.While they are in need of intensive care and hospitalized in the NICU, infants will receive conventional physiotherapy care three times a day. After discharge to the intermediate care unit (ICU), patients will receive care only once a day. Evaluations and interventions will be carried out five days a week (Monday to Friday), according to the logistics of the unit.
  Interventions: Procedure: Conventional Physiotherapy
- GP + hydrotherapy (GH) (Experimental): The sample will be evaluated once a day in the morning until they complete at least 11 intervention sessions of hydrotherapy in five moments: immediately before therapy, immediately after, 15, 30 and 60 minutes after the intervention. While they are in need of intensive care and hospitalized in the NICU, infants allocated to GH, hydrotherapy will be performed once a day, associated with two sessions of conventional physiotherapy. After discharge to the intermediate care unit (ICU), patients will receive care only once a day, both conventional physiotherapy and hydrotherapy. Evaluations and interventions will be carried out five days a week (Monday to Friday), according to the logistics of the unit.
  Interventions: Procedure: Hydrotherapy

INTERVENTIONS:
Procedure: Hydrotherapy — A re-sterilizable stainless steel bucket with an upper diameter of 30 cm, a depth of 32 cm, with water at a temperature between 37 and 38º Celsius will be used. The amount of water used will be sufficient to keep the baby submerged up to shoulder height. The baby will be immersed in the heated water of the bucket and will be suspended by occipital support performed by the physiotherapist, who alternates lateral-lateral and anteroposterior movements with only static suspension. The therapy will last from eight to ten minutes and will be discontinued if there is agitation, cyanosis, worsening respiratory distress or major evacuation. If the baby is using any type of ventilatory support or oxygen therapy, the same will be maintained during the procedure of hydrotherapy.
  Other Names: Hydrotherapies; Whirlpool Bath; Whirlpool Baths; Bath, Whirpool; Baths, Whirlpool
  Arms: GP + hydrotherapy (GH)
Procedure: Conventional Physiotherapy — Conventional physiotherapy consists of manipulations of Thoracoabdominal Rebalancing, a registered technique which uses simultaneous passive stretching of inspiratory muscles and stimulation of the diaphragm. The manipulation used to improve the dynamic diaphragm included the thoracic-abdominal and lower abdominal support maneuvers. Back repositioning was used to minimize posteriorization of the ribs and costal kyphosis due to thoracic distortion.
  Arms: Conventional physiotherapy (GP)

SUMMARY:
Premature newborns (PTNB) often develop bronchopulmonary dysplasia (BPD) which can be related to an inability to maintain differences in tonus patterns (extensor and flexor) between the cervical muscles, upper and lower limbs. Babies who develop BPD remain in the neonatal intensive care unit (NICU) for a prolonged period of time, undergoing a large number of painful procedures. Exposure to pain in premature newborns (PTNB) is one of the most damaging factors in the extrauterine environment, also causing stress, which can also interfere with tonus pattern. Therefore, the aim of this study is to evaluate the effects of hydrotherapy on muscular activity, pain, sleep and wakefulness, stress, physiological conditions and the need for oxygen in PTNB with BPD during hospitalization in the neonatal unit. EXPECTED RESULTS: Hydrotherapy is expected to relieve pain, improve sleep quality and reduce oxygen therapy and ventilatory support in hospitalized PTNB babies with BPD.

DETAILED DESCRIPTION:
INTRODUTION:The development of medicine in recent years, especially in neonatology, has contributed to a considerable reduction in mortality rates,however, with the increase in diseases that contribute to morbidity and mortality, such as bronchopulmonary dysplasia (BPD). Such condition is defined by the need for supplemental oxygen and/or ventilatory support for more than 28 days.One of the complications of BPD is the inability to maintain differences in tonus patterns(extensor and flexor) between the cervical muscles, upper and lower limbs, which can be assessed by surface electromyography (EMG). Babies who develop BPD remain in the neonatal intensive care unit (NICU) for a prolonged period of time, undergoing a large number of painful procedures.Exposure to pain in premature newborns (PTNB) is one of the most damaging factors in the extrauterine environment, also causing stress, which can be measured by salivary cortisol.Studies with pain relief methods in these babies are needed, such as hydrotherapy.This approach has proven to be effective and safe in reducing the signs of pain and stress and to improve sleep quality in preterm infants in the NICU, besides improving physiological parameters, such as peripheral oxygen saturation. OBJECTIVES: To evaluate the effects of hydrotherapy on muscular activity, pain, sleep and wakefulness, stress, physiological conditions and the need for oxygen in PTNB with BPD during hospitalization in the neonatal unit. METHODOLOGY: PTNB with a diagnosis of BPD will be randomized into two groups: conventional physiotherapy (GP) and conventional physiotherapy plus hydrotherapy (GH). The PTNB randomized to GH will be submitted to 11 hydrotherapy sessions. The PTNB from both groups will be submitted to evaluation of heart rate (HR), peripheral oxygen saturation (SpO2), respiratory rate (RR), pain, respiratory distress, sleep state, and wakefulness. The level of salivary cortisol and muscular activity (EMG) will also be evaluated. EXPECTED RESULTS: Hydrotherapy is expected to relieve pain, improve sleep quality and reduce oxygen therapy and ventilatory support in hospitalized PTNB babies with BPD.

ELIGIBILITY:
Inclusion Criteria:

* PTNB with gestational age less than 36 weeks with a diagnosis of BPD
* Babies without heart disease
* absence of central venous access, skin lesions, surgical wound, drainage and insufficiency of the adrenal gland.

Exclusion Criteria:

* Those unable to perform hydrotherapy for three consecutive days due to severe respiratory effort evaluated by the Silverman Andersen Bulletin and hemodynamic instability.

Ages: 23 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral oxygen saturation | Change from baseline peripheral oxygen saturation at 15, 30 and 60 minutes
  Peripheral oxygen saturation (%) will be measured using a pulse oximeter. Pulse oximetry is a method used to estimate the percentage of oxygen bound to hemoglobin in the blood and this variable will be assessed using a multi-parameter monitor.

SECONDARY OUTCOMES:
Pain evaluation | Change from baseline Neonatal Infant Pain Scale score at 15, 30 and 60 minutes.
  Evaluated by Neonatal Infant Pain Scale, scores ranging from 0 to 7.
State of sleep and wakefulness | Change from baseline Brazelton neonatal behavioral assessment scale scores at 15, 30 and 60 minutes.
  Neonatal behavioral assessed by Brazelton neonatal behavioral assessment scale, scores ranging from 1 to 6.
Breathing pattern | Change from baseline Silverman and Andersen bulletin scores at 15, 30 and 60 minutes.
  Respiratory distress assessed by Silverman and Andersen bulletin, scores ranging from 0 to 2.
Muscular activity | Change from baseline surface electromiography at 60 minutes.
  Muscular activity of trapezius, serratus anterior and erector spinae assessed by surface electromiography (Root Mean Square [RMS] in Volts).
Respiratory rate | Change from baseline respiratory rate at 15, 30 and 60 minutes.
  Respiratory rate (number of respiratory cycles per minute) will be assessed by a physiotherapist for one minute.
Heart rate | Change from baseline heart rate at 15, 30 and 60 minutes.
  Heart rate (number of heart beat per minute) will be assessed using a multi-parameter monitor.
Stress level | Change from baseline salivary cortisol at 30 minutes.
  Salivary cortisol (salivary cortisol in µg/dL) will be collected by aspirating saliva from the oral cavity of the infant with a 1mL syringe and depositing the contents in an appropriate storage container.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Probst, PhD, Principal Investigator — State University of Londrina
Locations (1):
- University Hospital, Londrina, Paraná, Brazil